CLINICAL TRIAL: NCT04984694
Title: Evaluation of Computerized Virtual Reality on FunctionalAbility and Quality of Life in Elderly
Brief Title: Computerized Virtual Reality in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MOST 105-2314-B-038 -063 -MY2
Record Dates: First submitted 2021-07-16; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2016-11

CONDITIONS: Cognitive Dysfunction; Cognitive Change; Independent Living; Quality of Life; Video Games
Keywords: cognitive dysfunction; computer-assisted instruction; independent living; video games; quality of life
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Parallel assignment A type of intervention model describing a clinical trial in which two or more groups of participants receive different interventions. For example, a three-arm parallel assignment involves three groups of participants. One group receives intervention (Computerized Virtual Reality program), one group receives social interaction, and the other group is the control group. So during the trial, participants in one group receive intervention "in parallel" to participants in the other group, who receive social interaction.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors were blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Computerized virtual reality training programs group (Hot-Plus group) (Experimental): Participants who are in Hot-Plus group will divide several small groups which will be 4 persons with mild cognitive impairment. Participants will receive computerized virtual reality training program by Hot-Plus as a group activity for one hour, once a week for 12 weeks.
  Interventions: Behavioral: Computerized virtual reality training programs group (Hot-Plus group)
- Social interaction group (Active Comparator): The participants in the social interaction group will come as a group for social interaction one hour weekly for 12 weeks.
  Interventions: Behavioral: Social interaction group
- Control group (No Intervention): The control group will maintain regular activities.

INTERVENTIONS:
Behavioral: Computerized virtual reality training programs group (Hot-Plus group) — In this study, the investigators utilised interactive-video games called "Xavix Hot Plus"(Hot-plus, Shinsedai[SSD] Co. Ltd, Shiga Japan), which was designed specifically for rehabilitation and reported high participant motivation and enjoyment while playing.
  Arms: Computerized virtual reality training programs group (Hot-Plus group)
Behavioral: Social interaction group — The social interaction group will get together as a group for social interaction one hour weekly for 12 weeks.
  Arms: Social interaction group

SUMMARY:
The number of dementia patients increased with aging population. People with subjective memory complaints or mild cognitive impairment (MCI) may have a high risk of developing dementia. Cognitive /memory training programs have shown the potential positive effects for improving or maintaining the cognitive progression. However, the impact of those cognitive progressions on functional ability and quality of life is not well understood. In addition, it appears to have large variability responsiveness among trained subjects. Most studies did not examine the individual difference associated with training. The major aim will evaluate the cognitive training programs on functional ability and quality of life in older adults. The results will be expected to understand the effectiveness of the computerized virtual reality training, improving or maintaining cognition, physical and psychosocial function, enhancing quality of life, and reducing the risk of developing disability even conversion into dementia in later life.

DETAILED DESCRIPTION:
Prevention strategies for dementia are needed because of the increasing prevalence of dementia. People with mild cognitive impairment are at high risk of developing a disability, even conversion into dementia in later life. Cognitive /memory training programs have shown the potential positive effects for improving or maintaining the cognitive progression. However, the impact of those cognitive progressions on functional ability and quality of life is not well understood. The major aim of this total project is to evaluate the short and long-term effects of computerized virtual reality training programs (Xavix Hot-Plus) on functional ability (cognition, physical and psychosocial function) and quality of life in older adults with mild cognitive impairment.

The experimental research design with three groups, one pretest and four posttests will be conducted to examine the short-term and long-term effects on cognition (primary outcome), physical (secondary outcome), psychosocial function (secondary outcome), and quality of life (secondary outcome). Independent adults will be recruited from the community base on sample criteria. The total subjects will be 160 to 190 older adults and the community care centers include all eligible participants will be randomly assigned into computerized virtual reality training programs group (Hot-Plus group) or social interaction group. The subjects for the control group will be recruited in the community and be referred by neurological, psychiatric, or gerontological physicians.

Participants who are in the Hot-Plus group will divide several small groups which will be 4 persons with mild cognitive impairment. Participants will receive a computerized virtual reality training program by Hot-Plus as a group activity one hour, once a week for 12 weeks. The participants in the social interaction group will come as a group for social interaction one hour weekly for 12 weeks. The control group will maintain their regular activities.

Data will be analysed by using SPSS version 18.0 (SPSS, Chicago, IL), with the significance level is set at p< .05. The normal distribution of the data will be evaluated using the Kolmogorov-Smirnov test. Mean, Standard deviation, frequency, and percentage will be performed to describe all variables. One-way analysis of variance (ANOVA) will be used to evaluate differences between groups according to the continuous variables, non-normal distribution of data will be calculated by Kruskasl-Wallis test. The chi-square test will be used for the comparison of categorical variables, and Fisher's exact test will be used due to the expected value less than four. Generalised Estimating Equation (GEE) will be used to examine the main effects, time effects, and interactions in outcomes over time.

The results will be expected to understand the effectiveness of the computerized virtual reality training, improving or maintaining cognition, physical, psychosocial function, enhancing quality of life, and reducing the risk of developing disability even conversion into dementia in later life.

ELIGIBILITY:
Inclusion Criteria:

* Equal to or older than 60 years old
* The SPMSQ scores range from 4-7 ( illiterate: 4-5, elementary: 5-6, junior high school: 6-7) or Clinical Dementia Rating Scale (CDR): 0.5
* Be able to communicate in Mandarin or Taiwanese
* Has the ability to see and hear well enough to follow the instructions
* Agree to participate in this study.

Exclusion Criteria:

* Activity restrictions from physician recommendation
* Unstable disease progress could affect their participation
* Surgery for joints or spinal cord within 6 months
* Unable to walk 50 meters with the assistant device
* Learning disability

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
Cognition-Global cognition | At baseline.
  Global cognition was measured by the Mini-Mental State Examination (MMSE), a modified version of a neuropsychological battery in the Consortium to Establish a Registry for Alzheimer's Disease (CERAD), which maximum score was 30 including orientation, memory, concentration, language, and praxis (Folstein, Folstein, & McHugh, 1975; Morris et al., 1989).
Cognition-Global cognition | Immediately after intervention.
  Global cognition was measured by the Mini-Mental State Examination (MMSE), a modified version of a neuropsychological battery in the Consortium to Establish a Registry for Alzheimer's Disease (CERAD), which maximum score was 30 including orientation, memory, concentration, language, and praxis (Folstein, Folstein, & McHugh, 1975; Morris et al., 1989).
Cognition-Global cognition | At 4 weeks after intervention.
  Global cognition was measured by the Mini-Mental State Examination (MMSE), a modified version of a neuropsychological battery in the Consortium to Establish a Registry for Alzheimer's Disease (CERAD), which maximum score was 30 including orientation, memory, concentration, language, and praxis (Folstein, Folstein, & McHugh, 1975; Morris et al., 1989).
Cognition-Global cognition | At 12 weeks after intervention.
  Global cognition was measured by the Mini-Mental State Examination (MMSE), a modified version of a neuropsychological battery in the Consortium to Establish a Registry for Alzheimer's Disease (CERAD), which maximum score was 30 including orientation, memory, concentration, language, and praxis (Folstein, Folstein, & McHugh, 1975; Morris et al., 1989).
Cognition-Global cognition | At 24 weeks after intervention.
  Global cognition was measured by the Mini-Mental State Examination (MMSE), a modified version of a neuropsychological battery in the Consortium to Establish a Registry for Alzheimer's Disease (CERAD), which maximum score was 30 including orientation, memory, concentration, language, and praxis (Folstein, Folstein, & McHugh, 1975; Morris et al., 1989).
Cognition-memory | At baseline.
  Memory was measured by the Word List test, contained three types as following (Morris et al., 1989; Welsh et al., 1994): 1) Immediately recall; 2) Delayed recall; 3) Recognition.
Cognition-memory | Immediately after intervention.
  Memory was measured by the Word List test, contained three types as following (Morris et al., 1989; Welsh et al., 1994): 1) Immediately recall; 2) Delayed recall; 3) Recognition.
Cognition-memory | At 4 weeks after intervention.
  Memory was measured by the Word List test, contained three types as following (Morris et al., 1989; Welsh et al., 1994): 1) Immediately recall; 2) Delayed recall; 3) Recognition.
Cognition-memory | At 12 weeks after intervention.
  Memory was measured by the Word List test, contained three types as following (Morris et al., 1989; Welsh et al., 1994): 1) Immediately recall; 2) Delayed recall; 3) Recognition.
Cognition-memory | At 24 weeks after intervention.
  Memory was measured by the Word List test, contained three types as following (Morris et al., 1989; Welsh et al., 1994): 1) Immediately recall; 2) Delayed recall; 3) Recognition.
Cognition-attention | At baseline.
  Attention was measured by the Digit Span (DS) subtest from the Taiwan version of the Wechsler Adult Intelligence Scale-Ⅲ (WAIS-IV; Wechsler, 2002), which contained two components: DS forward and DS backward.
Cognition-attention | Immediately after intervention.
  Attention was measured by the Digit Span (DS) subtest from the Taiwan version of the Wechsler Adult Intelligence Scale-Ⅲ (WAIS-IV; Wechsler, 2002), which contained two components: DS forward and DS backward.
Cognition-attention | At 4 weeks after intervention.
  Attention was measured by the Digit Span (DS) subtest from the Taiwan version of the Wechsler Adult Intelligence Scale-Ⅲ (WAIS-IV; Wechsler, 2002), which contained two components: DS forward and DS backward.
Cognition-attention | At 12 weeks after intervention.
  Attention was measured by the Digit Span (DS) subtest from the Taiwan version of the Wechsler Adult Intelligence Scale-Ⅲ (WAIS-IV; Wechsler, 2002), which contained two components: DS forward and DS backward.
Cognition-attention | At 24 weeks after intervention.
  Attention was measured by the Digit Span (DS) subtest from the Taiwan version of the Wechsler Adult Intelligence Scale-Ⅲ (WAIS-IV; Wechsler, 2002), which contained two components: DS forward and DS backward.
Cognition-visual/spatial function | At baseline.
  Visual/spatial function was measured by the Clock Drawing Test (CDT). Participants were asked to draw a clock face, place all the numbers on it, and set the time to 11 past 10 (Powlishta et al., 2002; Shulman, Shedletsky, & Silver, 1986).
Cognition-visual/spatial function | Immediately after intervention.
  Visual/spatial function was measured by the Clock Drawing Test (CDT). Participants were asked to draw a clock face, place all the numbers on it, and set the time to 11 past 10 (Powlishta et al., 2002; Shulman, Shedletsky, & Silver, 1986).
Cognition-visual/spatial function | At 4 weeks after intervention.
  Visual/spatial function was measured by the Clock Drawing Test (CDT). Participants were asked to draw a clock face, place all the numbers on it, and set the time to 11 past 10 (Powlishta et al., 2002; Shulman, Shedletsky, & Silver, 1986).
Cognition-visual/spatial function | At 12 weeks after intervention.
  Visual/spatial function was measured by the Clock Drawing Test (CDT). Participants were asked to draw a clock face, place all the numbers on it, and set the time to 11 past 10 (Powlishta et al., 2002; Shulman, Shedletsky, & Silver, 1986).
Cognition-visual/spatial function | At 24 weeks after intervention.
  Visual/spatial function was measured by the Clock Drawing Test (CDT). Participants were asked to draw a clock face, place all the numbers on it, and set the time to 11 past 10 (Powlishta et al., 2002; Shulman, Shedletsky, & Silver, 1986).
Cognition-executive function | At baseline.
  Executive function was measured by the Stroop Color and Word Test (SCWT)(Golden et al., 2002). It consisted of three subtasks: word reading (RED, GREEN, and BLUE), color naming (XXXX's colored in red, green, or blue ink), and incongruent color-word naming (the words RED, GREEN, and BLUE printed in not matching red, green, or blue ink).
Cognition-executive function | Immediately after intervention.
  Executive function was measured by the Stroop Color and Word Test (SCWT)(Golden et al., 2002). It consisted of three subtasks: word reading (RED, GREEN, and BLUE), color naming (XXXX's colored in red, green, or blue ink), and incongruent color-word naming (the words RED, GREEN, and BLUE printed in not matching red, green, or blue ink).
Cognition-executive function | At 4 weeks after intervention.
  Executive function was measured by the Stroop Color and Word Test (SCWT)(Golden et al., 2002). It consisted of three subtasks: word reading (RED, GREEN, and BLUE), color naming (XXXX's colored in red, green, or blue ink), and incongruent color-word naming (the words RED, GREEN, and BLUE printed in not matching red, green, or blue ink).
Cognition-executive function | At 12 weeks after intervention.
  Executive function was measured by the Stroop Color and Word Test (SCWT)(Golden et al., 2002). It consisted of three subtasks: word reading (RED, GREEN, and BLUE), color naming (XXXX's colored in red, green, or blue ink), and incongruent color-word naming (the words RED, GREEN, and BLUE printed in not matching red, green, or blue ink).
Cognition-executive function | At 24 weeks after intervention.
  Executive function was measured by the Stroop Color and Word Test (SCWT)(Golden et al., 2002). It consisted of three subtasks: word reading (RED, GREEN, and BLUE), color naming (XXXX's colored in red, green, or blue ink), and incongruent color-word naming (the words RED, GREEN, and BLUE printed in not matching red, green, or blue ink).

SECONDARY OUTCOMES:
Physical function-IADL | At baseline.
  Instrumental Activities of Daily Living (IADL) were evaluated with eight abilities, including shopping, transportation, meal preparation, ordinary housework, doing laundry, medications, phone use, and managing finances. Individual items are summed to produce a scale that ranges from 0 to 8 (Lawton, & Brody; 1969; Pashmdarfard & Azad, 2020).
Physical function-IADL | Immediately after intervention.
  IADL was evaluated with eight abilities including shopping, transportation, meal preparation, ordinary housework, doing laundry, medications, phone use, and managing finances. Individual items are summed to produce a scale that ranges from 0 to 8 (Lawton, & Brody; 1969; Pashmdarfard & Azad, 2020).
Physical function-IADL | At 4 weeks after intervention.
  IADL was evaluated with eight abilities including shopping, transportation, meal preparation, ordinary housework, doing laundry, medications, phone use, and managing finances. Individual items are summed to produce a scale that ranges from 0 to 8 (Lawton, & Brody; 1969; Pashmdarfard & Azad, 2020).
Physical function-IADL | At 12 weeks after intervention.
  IADL was evaluated with eight abilities including shopping, transportation, meal preparation, ordinary housework, doing laundry, medications, phone use, and managing finances. Individual items are summed to produce a scale that ranges from 0 to 8 (Lawton, & Brody; 1969; Pashmdarfard & Azad, 2020).
Physical function-IADL | At 24 weeks after intervention.
  IADL was evaluated with eight abilities including shopping, transportation, meal preparation, ordinary housework, doing laundry, medications, phone use, and managing finances. Individual items are summed to produce a scale that ranges from 0 to 8 (Lawton, & Brody; 1969; Pashmdarfard & Azad, 2020).
Physical function-senior fitness test (SFT) | At baseline.
  A series of functional test include chair stand test, 8-ft up and go test, chair sit and reach test, 6-min walk test, and unipedal stance test was developed by Rikli & Jones.
  It has good reliability and validity and test-retest reliability is above 0.9 (Rikli & Jones, 2001).
Physical function-senior fitness test (SFT) | Immediately after intervention.
  A series of functional test include chair stand test, 8-ft up and go test, chair sit and reach test, 6-min walk test, and unipedal stance test was developed by Rikli & Jones.
  It has good reliability and validity and test-retest reliability is above 0.9 (Rikli & Jones, 2001).
Physical function-senior fitness test (SFT) | At 4 weeks after intervention.
  A series of functional test include chair stand test, 8-ft up and go test, chair sit and reach test, 6-min walk test, and unipedal stance test was developed by Rikli & Jones.
  It has good reliability and validity and test-retest reliability is above 0.9 (Rikli & Jones, 2001).
Physical function-senior fitness test (SFT) | At 12 weeks after intervention.
  A series of functional test include chair stand test, 8-ft up and go test, chair sit and reach test, 6-min walk test, and unipedal stance test was developed by Rikli & Jones.
  It has good reliability and validity and test-retest reliability is above 0.9 (Rikli & Jones, 2001).
Physical function-senior fitness test (SFT) | At 24 weeks after intervention.
  A series of functional test include chair stand test, 8-ft up and go test, chair sit and reach test, 6-min walk test, and unipedal stance test was developed by Rikli & Jones.
  It has good reliability and validity and test-retest reliability is above 0.9 (Rikli & Jones, 2001).
Physical function-unipedal stance test (UST) | At baseline.
  Unipedal stance test was used to examine the static balance on the preferred leg. Participants performed three trials with the eyes open during the test (Goldberg, Casby, & Wasielewski, 2011) .
Physical function-unipedal stance test (UST) | Immediately after intervention.
  Unipedal stance test was used to examine the static balance on the preferred leg. Participants performed three trials with the eyes open during the test (Goldberg, Casby, & Wasielewski, 2011) .
Physical function-unipedal stance test (UST) | At 4 weeks after intervention.
  Unipedal stance test was used to examine the static balance on the preferred leg. Participants performed three trials with the eyes open during the test (Goldberg, Casby, & Wasielewski, 2011) .
Physical function-unipedal stance test (UST) | At 12 weeks after intervention.
  Unipedal stance test was used to examine the static balance on the preferred leg. Participants performed three trials with the eyes open during the test (Goldberg, Casby, & Wasielewski, 2011) .
Physical function-unipedal stance test (UST) | At 24 weeks after intervention.
  Unipedal stance test was used to examine the static balance on the preferred leg. Participants performed three trials with the eyes open during the test (Goldberg, Casby, & Wasielewski, 2011) .
Psychosocial factors-Global Well-Being Scale (GWBS) | At baseline.
  Global Well-Being Scale (GWBS): It is a 10-centimeter visual analog scale to measures individuals' perception of well-being. The score of GWBS ranged from 0 to 10 (Hawk et al., 2010).
  Analog Scale (VAS) with a ten-centimeter horizontal line (Hawk et al., 2010).
Psychosocial factors-Global Well-Being Scale (GWBS) | Immediately after intervention.
  Global Well-Being Scale (GWBS): It is a 10-centimeter visual analog scale to measures individuals' perception of well-being. The score of GWBS ranged from 0 to 10 (Hawk et al., 2010).
  Analog Scale (VAS) with a ten-centimeter horizontal line (Hawk et al., 2010).
Psychosocial factors-Global Well-Being Scale (GWBS) | At 4 weeks after intervention.
  Global Well-Being Scale (GWBS): It is a 10-centimeter visual analog scale to measures individuals' perception of well-being. The score of GWBS ranged from 0 to 10 (Hawk et al., 2010).
  Analog Scale (VAS) with a ten-centimeter horizontal line (Hawk et al., 2010).
Psychosocial factors-Global Well-Being Scale (GWBS) | At 12 weeks after intervention.
  Global Well-Being Scale (GWBS): It is a 10-centimeter visual analog scale to measures individuals' perception of well-being. The score of GWBS ranged from 0 to 10 (Hawk et al., 2010).
  Analog Scale (VAS) with a ten-centimeter horizontal line (Hawk et al., 2010).
Psychosocial factors-Global Well-Being Scale (GWBS) | At 24 weeks after intervention.
  Global Well-Being Scale (GWBS): It is a 10-centimeter visual analog scale to measures individuals' perception of well-being. The score of GWBS ranged from 0 to 10 (Hawk et al., 2010).
  Analog Scale (VAS) with a ten-centimeter horizontal line (Hawk et al., 2010).
Psychosocial factors-Interpersonal Relationship Scale (IRS) | At baseline.
  This scale was developed by Chang and Su (2011) in order to know the interpersonal relationship for middle-aged and older Adults.
  It's composed of 22 questions related to the interpersonal relationship: close interaction, approach to others, and friendship support (Chang & Su, 2011).
Psychosocial factors-Interpersonal Relationship Scale (IRS) | Immediately after intervention.
  This scale was developed by Chang and Su (2011) in order to know the interpersonal relationship for middle-aged and older Adults.
  It's composed of 22 questions related to the interpersonal relationship: close interaction, approach to others, and friendship support (Chang & Su, 2011).
Psychosocial factors-Interpersonal Relationship Scale (IRS) | At 4 weeks after intervention.
  This scale was developed by Chang and Su (2011) in order to know the interpersonal relationship for middle-aged and older Adults.
  It's composed of 22 questions related to the interpersonal relationship: close interaction, approach to others, and friendship support (Chang & Su, 2011).
Psychosocial factors-Interpersonal Relationship Scale (IRS) | At 12 weeks after intervention.
  This scale was developed by Chang and Su (2011) in order to know the interpersonal relationship for middle-aged and older Adults.
  It's composed of 22 questions related to the interpersonal relationship: close interaction, approach to others, and friendship support (Chang & Su, 2011).
Psychosocial factors-Interpersonal Relationship Scale (IRS) | At 24 weeks after intervention.
  This scale was developed by Chang and Su (2011) in order to know the interpersonal relationship for middle-aged and older Adults.
  It's composed of 22 questions related to the interpersonal relationship: close interaction, approach to others, and friendship support (Chang & Su, 2011).
Psychosocial factors-Geriatric Depression Scale-Short Form (GDS-SF) | At baseline.
  Chinese version of the GDS-S consisted 15 items with yes/no questions and higher scores indicate a more severe level of depression (Lu, Liu, & Yu, 1998; Pfeiffer, 1975).
Psychosocial factors-Geriatric Depression Scale-Short Form (GDS-SF) | Immediately after intervention.
  Chinese version of the GDS-S consisted 15 items with yes/no questions and higher scores indicate a more severe level of depression (Lu, Liu, & Yu, 1998; Pfeiffer, 1975).
Psychosocial factors-Geriatric Depression Scale-Short Form (GDS-SF) | At 4 weeks after intervention.
  Chinese version of the GDS-S consisted 15 items with yes/no questions and higher scores indicate a more severe level of depression (Lu, Liu, & Yu, 1998; Pfeiffer, 1975).
Psychosocial factors-Geriatric Depression Scale-Short Form (GDS-SF) | At 12 weeks after intervention.
  Chinese version of the GDS-S consisted 15 items with yes/no questions and higher scores indicate a more severe level of depression (Lu, Liu, & Yu, 1998; Pfeiffer, 1975).
Psychosocial factors-Geriatric Depression Scale-Short Form (GDS-SF) | At 24 weeks after intervention.
  Chinese version of the GDS-S consisted 15 items with yes/no questions and higher scores indicate a more severe level of depression (Lu, Liu, & Yu, 1998; Pfeiffer, 1975).
Quality of Life-EQ5D-Utility | At baseline.
  EQ-5D-3L Taiwanese version questionnaire was selected to measure health-related quality of life (HRQOL) which was recommended in older adults and people with mild dementia (Aguirre, Kang, Hoare, Edwards, & Orrell, 2016; León-Salas et al., 2015). According to the self-report index scores, it can be converted to a single summary utility score by using the time trade-off (TTO) technique. The range of this EQ-5D-3L utility score (EQ5D-Utility) was -0.67 to 1.00 by using the Taiwanese value set (Lee et al., 2013), as the score closer to 1 indicated the better health, a negative score indicated worse than dead, and a 0.5 score could be acceptable.
Quality of Life-EQ5D-Utility | Immediately after intervention.
  EQ-5D-3L Taiwanese version questionnaire was selected to measure health-related quality of life (HRQOL) which was recommended in older adults and people with mild dementia (Aguirre, Kang, Hoare, Edwards, & Orrell, 2016; León-Salas et al., 2015). According to the self-report index scores, it can be converted to a single summary utility score by using the time trade-off (TTO) technique. The range of this EQ-5D-3L utility score (EQ5D-Utility) was -0.67 to 1.00 by using the Taiwanese value set (Lee et al., 2013), as the score closer to 1 indicated the better health, a negative score indicated worse than dead, and a 0.5 score could be acceptable.
Quality of Life-EQ5D-Utility | At 4 weeks after intervention.
  EQ-5D-3L Taiwanese version questionnaire was selected to measure health-related quality of life (HRQOL) which was recommended in older adults and people with mild dementia (Aguirre, Kang, Hoare, Edwards, & Orrell, 2016; León-Salas et al., 2015). According to the self-report index scores, it can be converted to a single summary utility score by using the time trade-off (TTO) technique. The range of this EQ-5D-3L utility score (EQ5D-Utility) was -0.67 to 1.00 by using the Taiwanese value set (Lee et al., 2013), as the score closer to 1 indicated the better health, a negative score indicated worse than dead, and a 0.5 score could be acceptable.
Quality of Life-EQ5D-Utility | At 12 weeks after intervention.
  EQ-5D-3L Taiwanese version questionnaire was selected to measure health-related quality of life (HRQOL) which was recommended in older adults and people with mild dementia (Aguirre, Kang, Hoare, Edwards, & Orrell, 2016; León-Salas et al., 2015). According to the self-report index scores, it can be converted to a single summary utility score by using the time trade-off (TTO) technique. The range of this EQ-5D-3L utility score (EQ5D-Utility) was -0.67 to 1.00 by using the Taiwanese value set (Lee et al., 2013), as the score closer to 1 indicated the better health, a negative score indicated worse than dead, and a 0.5 score could be acceptable.
Quality of Life-EQ5D-Utility | At 24 weeks after intervention.
  EQ-5D-3L Taiwanese version questionnaire was selected to measure health-related quality of life (HRQOL) which was recommended in older adults and people with mild dementia (Aguirre, Kang, Hoare, Edwards, & Orrell, 2016; León-Salas et al., 2015). According to the self-report index scores, it can be converted to a single summary utility score by using the time trade-off (TTO) technique. The range of this EQ-5D-3L utility score (EQ5D-Utility) was -0.67 to 1.00 by using the Taiwanese value set (Lee et al., 2013), as the score closer to 1 indicated the better health, a negative score indicated worse than dead, and a 0.5 score could be acceptable.
Quality of Life-EQ5D-visual analogue scale | At baseline.
  A 20-cm visual analogue scale in which respondents are asked to rate their current health status ranging from 0 (Worst imaginable health state) to 100 (Chang et al., 2007; EuroQol Research Foundation, 2018).
Quality of Life-EQ5D-visual analogue scale | Immediately after intervention.
  A 20-cm visual analogue scale in which respondents are asked to rate their current health status ranging from 0 (Worst imaginable health state) to 100 (Chang et al., 2007; EuroQol Research Foundation, 2018).
Quality of Life-EQ5D-visual analogue scale | At 4 weeks after intervention.
  A 20-cm visual analogue scale in which respondents are asked to rate their current health status ranging from 0 (Worst imaginable health state) to 100 (Chang et al., 2007; EuroQol Research Foundation, 2018).
Quality of Life-EQ5D-visual analogue scale | At 12 weeks after intervention.
  A 20-cm visual analogue scale in which respondents are asked to rate their current health status ranging from 0 (Worst imaginable health state) to 100 (Chang et al., 2007; EuroQol Research Foundation, 2018).
Quality of Life-EQ5D-visual analogue scale | At 24 weeks after intervention.
  A 20-cm visual analogue scale in which respondents are asked to rate their current health status ranging from 0 (Worst imaginable health state) to 100 (Chang et al., 2007; EuroQol Research Foundation, 2018).

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Chi Chang, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- TMU-Shuang-Ho Hospital, Taipei Medical University, New Taipei City, Taiwan

REFERENCES:
- [Background] Supreme Investment. Interactive health service system. Supreme Investment website. https://supremeinvest.co/hotplus/. Updated 2016. Accessed March 17, 2017.
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Morris JC, Heyman A, Mohs RC, Hughes JP, van Belle G, Fillenbaum G, Mellits ED, Clark C. The Consortium to Establish a Registry for Alzheimer's Disease (CERAD). Part I. Clinical and neuropsychological assessment of Alzheimer's disease. Neurology. 1989 Sep;39(9):1159-65. doi: 10.1212/wnl.39.9.1159. PMID 2771064
- [Background] Welsh KA, Butters N, Mohs RC, Beekly D, Edland S, Fillenbaum G, Heyman A. The Consortium to Establish a Registry for Alzheimer's Disease (CERAD). Part V. A normative study of the neuropsychological battery. Neurology. 1994 Apr;44(4):609-14. doi: 10.1212/wnl.44.4.609. PMID 8164812
- [Background] Powlishta KK, Von Dras DD, Stanford A, Carr DB, Tsering C, Miller JP, Morris JC. The clock drawing test is a poor screen for very mild dementia. Neurology. 2002 Sep 24;59(6):898-903. doi: 10.1212/wnl.59.6.898. PMID 12297574
- [Background] Shulman K, Shedletsky R, Silver I. The challenge of time: Clock-drawing and cognitive function in the elderly. Int J Geriat Psychiatry. 1986:1(2):135-140.
- [Background] Golden CJ. A group version of the Stroop Color and Word Test. J Pers Assess. 1975 Aug;39(4):386-8. doi: 10.1207/s15327752jpa3904_10. PMID 16367401
- [Background] Pashmdarfard M, Azad A. Assessment tools to evaluate Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) in older adults: A systematic review. Med J Islam Repub Iran. 2020 Apr 13;34:33. doi: 10.34171/mjiri.34.33. eCollection 2020. PMID 32617272
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Rikli RE, Jones CJ. Senior Fitness Test Manual. Champaign: Human Kinetics; 2001.
- [Background] Hawk C, Dusio ME, Wallace H, Bernard T, Rexroth C. Development of a patient-centered instrument for the assessment of global well-being: a study of reliability, validity, and clinical responsiveness. Palmer J Res. 1995;2(1):15-22.
- [Background] Chang W J, Su MP. Exploring the effects of self-concept and interpersonal relationship who attends the music program for middle-aged and elderly adults in community. Journal of Community Research. 2011:2:109-157.
- [Background] Liu HC, Fuh JL, Wang SJ, Liu CY, Larson EB, Lin KN, Wang HC, Chou P, Wu ZA, Lin CH, Wang PN, Teng EL. Prevalence and subtypes of dementia in a rural Chinese population. Alzheimer Dis Assoc Disord. 1998 Sep;12(3):127-34. doi: 10.1097/00002093-199809000-00002. PMID 9772013
- [Background] Pfeiffer E. A short portable mental status questionnaire for the assessment of organic brain deficit in elderly patients. J Am Geriatr Soc. 1975 Oct;23(10):433-41. doi: 10.1111/j.1532-5415.1975.tb00927.x. PMID 1159263
- [Background] Lee HY, Hung MC, Hu FC, Chang YY, Hsieh CL, Wang JD. Estimating quality weights for EQ-5D (EuroQol-5 dimensions) health states with the time trade-off method in Taiwan. J Formos Med Assoc. 2013 Nov;112(11):699-706. doi: 10.1016/j.jfma.2012.12.015. Epub 2013 Feb 12. PMID 24183199
- [Background] Chang TJ, Tarn YH, Hsieh CL, Liou WS, Shaw JW, Chiou XG. Taiwanese version of the EQ-5D: validation in a representative sample of the Taiwanese population. J Formos Med Assoc. 2007 Dec;106(12):1023-31. doi: 10.1016/S0929-6646(08)60078-9. PMID 18194908
- [Background] EuroQol Research Foundation. EQ-5D-3L User Guidet, 2018. https://euroqol.org/publications/user-guides/. Updated October, 2018. Accessed August 16, 2019.